CLINICAL TRIAL: NCT00867321
Title: Phase I/II Randomized Trial of Sorafenib and Bevacizumab as First-Line Therapy in Patients With Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Bevacizumab and Sorafenib as First-Line Therapy in Treating Patients With Locally Advanced or Metastatic Liver Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0745; NCI-2009-01178 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000637866 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Bevacizumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Phase II) (Experimental): Patients receive oral sorafenib tosylate on days 1-28 twice daily and bevacizumab IV on days 1 and 15.
  Interventions: Biological: bevacizumab; Drug: sorafenib tosylate
- Arm II (Phase II) (Experimental): Patients receive oral sorafenib tosylate twice daily on days 1-28.
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Arms: Arm I (Phase II)
Drug: sorafenib tosylate — Given orally

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab and sorafenib may also stop the growth of liver cancer by blocking blood flow to the tumor.

PURPOSE: This randomized phase I/II trial is studying the best dose of bevacizumab when given together with sorafenib as first-line therapy in treating patients with locally advanced or metastatic liver cancer.(Phase I closed to accrual as of 11/03/2010)

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of bevacizumab in combination with sorafenib tosylate in patients with locally advanced or metastatic hepatocellular carcinoma. (Phase I closed to accrual as of 11/03/2010)
* Determine time to progression in these patients. (Phase II)

Secondary

* Determine the safety of this regimen in these patients. (Phase I closed to accrual as of 11/03/2010)
* Assess tolerability of this regimen in these patients. (Phase I closed to accrual as of 11/03/2010)
* Determine overall survival of these patients. (Phase II)
* Determine tumor response (at 6 months) in patients treated with this regimen. (Phase II)
* Determine progression-free survival of these patients. (Phase II)
* Determine response rate in patients treated with this regimen. (Phase II)
* Assess the occurrence of adverse events in these patients. (Phase II)

Tertiary

* Determine the relationship between tumor biomarkers and circulating biomarkers of vascular response and clinical outcome in patients treated with this regimen.

OUTLINE: This is a phase I, dose escalation study followed by a randomized phase II study.

* Phase I (closed to accrual as of 11/03/2010): Patients receive oral sorafenib tosylate twice daily on days 1-28 and bevacizumab IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients are stratified according to gender (female vs male), ECOG performance status (0 vs 1), and Child-Pugh class (A vs B7). Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral sorafenib tosylate on days 1-28 twice daily and bevacizumab IV on days 1 and 15.
  * Arm II: Patients receive oral sorafenib tosylate twice daily on days 1-28. In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for analysis of circulating endothelial cells and circulating endothelial progenitor cells and angiogenic proteins in plasma by ELISA.

After completion of study treatment, patients are followed for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma

  * Locally advanced or metastatic disease that is not amenable to treatment with surgery or to orthotopic liver transplant
  * Child Pugh class A or B7 disease
* Measurable disease
* No mixed cholangiocarcinoma/hepatocellular carcinoma
* No current or previously resected brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* ANC ≥ 1,200/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 5 times ULN
* Alkaline phosphatase ≤ 5 times ULN
* Urine protein ≤ 1+ by urine protein:creatinine ratio OR 24-hour urine protein < 1 g
* QTc interval ≤ 500 msec on baseline EKG
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 2 weeks after sorafenib tosylate and 6 months after bevacizumab
* None of the following risk factors for decreased LVEF:

  * Prior treatment with anthracyclines
  * History of myocardial infarction within the past 12 months
* No uncontrolled hypertension (defined as systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 100 mm Hg) despite optimal medical management
* No New York Heart Association class III-IV congestive heart failure
* No cardiac ventricular arrhythmias requiring antiarrhythmic therapy
* No history of hypertensive crisis or hypertensive encephalopathy
* No cardiac ventricular arrhythmia requiring anti-arrhythmic therapy within the past 6 months
* None of the following within the past 6 months:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina or angina
  * Clinically significant peripheral artery disease (i.e., claudication in less than one block) or any other arterial thrombotic event
  * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess
  * Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis
* No active or recent history of hemoptysis (≥ ½ teaspoon of bright red blood per episode) within the past 30 days
* No evidence of bleeding diathesis (greater than normal risk of bleeding) or coagulopathy (in the absence of therapeutic anticoagulation)
* No significant traumatic injury within the past 4 weeks
* No serious or non-healing wound, ulcer, or bone fracture
* No uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* No other active malignancy within the past 3 years, except nonmelanotic skin cancer or carcinoma in situ of the cervix
* No comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab or sorafenib tosylate

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy regimens for hepatocellular carcinoma
* No prior external beam radiation to the primary site
* No prior central thoracic radiation therapy (RT), including RT to the heart
* No prior radiation (if given for another malignancy) to ≥ 25% of the bone marrow
* At least 6 weeks since prior chemoembolization, radioembolization, radiofrequency ablation, or other local ablative therapies
* More than 4 weeks since prior biologic, hormonal, or immune therapy
* More than 4 weeks since prior and no concurrent major surgical procedure or open biopsy
* More than 7 days since prior core biopsy or other minor surgical procedure (placement of a vascular access device allowed)
* No concurrent investigational agent which would be considered as a treatment for the primary neoplasm
* No concurrent anticoagulants, except low-dose warfarin or heparin for deep venous thrombosis prophylaxis
* No other concurrent treatment for prior malignancy (other than hormonal therapy)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (177):
- United States (177):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Bettendorf, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Hubbard JM, Mahoney MR, Loui WS, Roberts LR, Smyrk TC, Gatalica Z, Borad M, Kumar S, Alberts SR. Phase I/II Randomized Trial of Sorafenib and Bevacizumab as First-Line Therapy in Patients with Locally Advanced or Metastatic Hepatocellular Carcinoma: North Central Cancer Treatment Group Trial N0745 (Alliance). Target Oncol. 2017 Apr;12(2):201-209. doi: 10.1007/s11523-016-0467-0. PMID 27943153

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level 0: Patients receive:> > Oral 400 mg BID Sorafenib on days 1-28.>
  > 1.25 mg/kg Bevacizumab IV on days 1, 15.
- Phase I: Dose Level -1: Patients receive:> > Oral 400 mg BID Sorafenib, 5 consecutive days out of each 7 days>
  > 1.25 mg/kg Bevacizumab IV on days 1, 15
- Phase I: Dose Level -2a: Patients receive:> > Oral 200 mg BID Sorafenib days 1-28>
  > 2.5 mg/kg Bevacizumab IV on days 1, 15
- Phase I: Dose Level -2: Patients receive:> > Oral 200 mg BID Sorafenib days 1-28>
  > 1.25 mg/kg Bevacizumab IV on days 1, 15
Period: Overall Study
Arm/Group | Arm I (Phase II) | Arm II (Phase II) | Phase I: Dose Level 0 | Phase I: Dose Level -1 | Phase I: Dose Level -2a | Phase I: Dose Level -2
Started | 4 | 3 | 3 | 6 | 5 | 3
Completed | 4 | 2 | 3 | 6 | 5 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients were used to analyze baseline characteristics.
Groups:
- All Phase I Patients: This includes all patients who participated in the phase I dose escalation portion of the trial.
- Total: Total of all reporting groups
Arm/Group | Arm I (Phase II) | Arm II (Phase II) | All Phase I Patients | Total
Number analyzed (Participants) | 4 | 3 | 17 | 24
Age, Continuous [Median (Full Range); unit: years] | 58.5 [54 to 80] | 55 [52 to 61] | 66 [18 to 79] | 60.5 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5
  Male | 3 | 2 | 14 | 19
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 17 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Phase I)
Description: MTD is defined as the dose level below the lowest dose that induces dose limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients). If dose level (-1) is not tolerable, but dose (-3) or (-2) is below or at MTD, testing of alternate dose levels (-2a, -3a, -3b) will occur as outlined in the table. The number of dose limiting toxicities will be reported here.
Time Frame: From baseline up to 3 years post treatment
Population: All eligible patients were treated and analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Dose Level 0: Patients receive:
  >
  > Oral 400 mg BID Sorafenib on days 1-28.
  >
  > 1.25 mg/kg Bevacizumab IV on days 1, 15.
- Phase I: Dose Level -1: Patients receive:
  >
  > Oral 400 mg BID Sorafenib, 5 consecutive days out of each 7 days
  >
  > 1.25 mg/kg Bevacizumab IV on days 1, 15
- Phase I: Dose Level -2a (Maximum Tolerated Dose): Patients receive:
  >
  > Oral 200 mg BID Sorafenib days 1-28
  >
  > 2.5 mg/kg Bevacizumab IV on days 1, 15
- Phase I: Dose Level -2: Patients receive:
  >
  > Oral 200 mg BID Sorafenib days 1-28
  >
  > 1.25 mg/kg Bevacizumab IV on days 1, 15
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level -1 | Phase I: Dose Level -2a (Maximum Tolerated Dose) | Phase I: Dose Level -2
Number analyzed (Participants) | 3 | 6 | 5 | 3
Participants | 2 | 3 | 0 | 0

2. Primary Outcome: Time to Progression (TTP) (Phase II)
Description: Time to progression is defined to be the length of time from study registration to a) date of disease progression as defined by section 11.0, or b) last follow-up. If a patient dies without documentation of disease progression, the patient will be considered to have had a tumor progression at the time of death unless there is sufficient documented evidence to conclude no progression occurred prior to death. Kaplan-Meier survival curves will be used to estimate the distribution of TTP.
Time Frame: From baseline up to 3 years post treatment
Population: 6 of 7 patients have had at least one post-baseline assessment of disease and were used for this endpoint.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I (Phase II) | Arm II (Phase II)
Number analyzed (Participants) | 4 | 2
years | 8.6 [.4 to 16.3] | 13.3 [4.4 to NA] — The upper confidence bound was non-estimable.

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the length of time from date of registration to a) date of death due to any cause or b) last follow-up. Kaplan-Meier survival curves will be used to estimate the distribution of OS.
Time Frame: Up to 3 years post treatment
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Patients: Due to lack of accrual Overall Survival was estimated using all patients
Arm/Group | All Patients
Number analyzed (Participants) | 6
Months | 13.3 [4.4 to NA] — Upper confidence interval was not reached

4. Secondary Outcome: Tumor Response at 6 Months
Description: Tumor response (at 6 months) is defined as the number of responses (complete or partial response per Section 11) over the number of eligible patients observed for at least 6 months. Tumor response will be evaluated using simple estimates of proportions.
Time Frame: 6 months
Population: No patients were analyzed for this endpoint because data was not collected for it
Arm/Group | Arm I (Phase II) | Arm II (Phase II)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Phase I: Dose Level 0: Patients receive:
  Oral 400 mg BID Sorafenib on days 1-28.
  1.25 mg/kg Bevacizumab IV on days 1, 15
- Phase I: Dose Level -1: Patients receive:
  Oral 400 mg BID Sorafenib, 5 consecutive days out of each 7 days
  1.25 mg/kg Bevacizumab IV on days 1, 15
- Phase I: Dose Level -2a: Patients receive:
  Oral 200 mg BID Sorafenib days 1-28
  2.5 mg/kg Bevacizumab IV on days 1, 15
- Phase I: Dose Level -2: Patients receive:
  Oral 200 mg BID Sorafenib days 1-28
  1.25 mg/kg Bevacizumab IV on days 1, 15
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level -1 | Phase I: Dose Level -2a | Phase I: Dose Level -2 | Arm I (Phase II) | Arm II (Phase II)
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 0/5 | 0/3 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 5/5 | 3/3 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 0 (N=3) | Phase I: Dose Level -1 (N=6) | Phase I: Dose Level -2a (N=5) | Phase I: Dose Level -2 (N=3) | Arm I (Phase II) (N=4) | Arm II (Phase II) (N=3)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 0 (N=3) | Phase I: Dose Level -1 (N=6) | Phase I: Dose Level -2a (N=5) | Phase I: Dose Level -2 (N=3) | Arm I (Phase II) (N=4) | Arm II (Phase II) (N=3)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorder (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (7) | 1 (1) | 1 (10) | 1 (1) | 2 (16)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Fatigue (General disorders) | 3 (7) | 6 (14) | 4 (20) | 3 (8) | 4 (11) | 3 (15)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (3)
Bilirubin increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (7)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Leukocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (7) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (12) | 2 (14) | 2 (6) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (7)
Hypertension (Vascular disorders) | 2 (3) | 1 (2) | 1 (1) | 1 (2) | 4 (8) | 3 (6)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less